CLINICAL TRIAL: NCT01766999
Title: Methemoglobinemia After Liposuction Under Tumescent Local Anesthesia - Timecourse and Diagnostics by Pulse Oximetry and Blood Gas Analysis.
Brief Title: Methemoglobinemia After Liposuction - Diagnostic by Pulse Oximetry and Blood Gas Analysis.
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Hartmut Gehring, Prof. Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: MetHb02
Record Dates: First submitted 2013-01-04; First posted 2013-01-11 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Methemoglobinemia
Keywords: pulse oximetry; tumescent anesthesia
MeSH Terms: conditions — Methemoglobinemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpMetHb > 8%: hemoximetric MetHb measurements triggered

SUMMARY:
Tumescent local anesthesia is a procedure which is frequently performed for plastic cosmetic surgical procedures such as liposuction. The subcutaneous adipose tissue is infiltrated with large volumes of a solution which also contain local anesthetics. However local anesthetics, can also lead to a marked production of methemoglobin. New generation pulse oximeters are able to measure SpMetHb non-invasivly.

The aim of this study is:

1. to investigate multi-wavelength pulse oximetry as a monitoring method for patients at increased risk for methemoglobinemia.
2. to illustrate MetHb concentrations over a course of 24 hours after a liposuction employing tumescent anesthesia has been carried out.

ELIGIBILITY:
Inclusion Criteria:

* planned liposuction in tumescent local anesthesia

Exclusion Criteria:

* hematologic disorders

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - female patients scheduled for liposuction
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Correlation between hemoximetric and pulseoximetric measured methemoglobin | 24 hours

SECONDARY OUTCOMES:
Time course of MetHb concentration following liposuction employing tumescent anesthesia. | 24 hours